CLINICAL TRIAL: NCT06459934
Title: Clinical Outcomes of Cardiovascular Disease: a Prospective Cohort Study
Brief Title: Clinical Outcomes of Cardiovascular Disease
Acronym: CLEAR
Status: Recruiting | Type: Observational
Sponsor: Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Xiang Xie, Director, Xinjiang Medical University
Other Study IDs: 20240606
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Cardiovascular Diseases; Heart Failure; Coronary Artery Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collect 5ml of fasting blood and store at -80 ℃.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a prospective, single center cohort study that primarily registers the clinical characteristics, outcomes, and influencing factors of patients with different types of cardiovascular diseases. Evaluate multiple examination indicators of patients at baseline, 1 year and longer, and follow up on the incidence of major cardiovascular and cerebrovascular adverse events, heart failure readmission, death, and other endpoint events.

DETAILED DESCRIPTION:
This study is a prospective, single center cohort study that primarily registers the clinical characteristics, outcomes, and influencing factors of patients with different types of cardiovascular diseases. Mainly including coronary heart disease, cardiomyopathy, hypertension, heart failure and other diseases, multiple examination indicators are evaluated for patients at baseline, 1 year and longer periods of time. The primary endpoints for coronary heart disease are all-cause mortality, cardiogenic death, non fatal myocardial infarction, hospitalization for heart failure, and major cardiovascular adverse events. The primary endpoints for cardiomyopathy are all-cause mortality, cardiogenic death, hospitalization for heart failure, and major cardiovascular adverse events. The primary endpoints for hypertension are stroke, all-cause mortality, cardiogenic death, hospitalization for heart failure, and major cardiovascular and cerebrovascular adverse events. The primary endpoints for heart failure are all-cause mortality, cardiogenic death, readmission for heart failure, and major cardiovascular adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Coronary heart disease According to coronary angiography and coronary CTA, at least one coronary artery has a degree of stenosis greater than 50%.
2. Hypertension Hypertension is defined as office systolic blood pressure is ≥ 140mmHg and/or the diastolic blood pressure is ≥ 90mmHg without the use of antihypertensive drugs.
3. Heart failure There is a clear history of organic heart disease, clinical symptoms and signs of heart failure, and objective evidence of heart failure.
4. Cardiomyopathy Including defined dilated cardiomyopathy, hypertrophic cardiomyopathy, restrictive cardiomyopathy, etc.
5. Able to sign informed consent form.

Exclusion Criteria:

1. Age<18 years old, or>80 years old.
2. Patients with various malignant tumors.
3. Liver dysfunction (defined as ALT or total bilirubin greater than three times the upper normal limit).
4. Renal insufficiency (defined as blood creatinine exceeding 1.5 times the upper normal limit).
5. Those who have participated in other clinical studies within the past three months.
6. Individuals without legal capacity or with limited legal capacity.
7. Any situation where the researcher deems it unsuitable to participate in the clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population mainly includes patients with different types of cardiovascular diseases. Mainly including coronary heart disease, cardiomyopathy, hypertension, heart failure and other diseases.
Sampling Method: Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
All cause death | 1 year.
  Death caused by various reasons.
Cardiac death | 1 year.
  Death caused by cardiac reasons.
Main adverse cardiovascular events（MACE） | 1 year.
  The composite endpoint for hospitalization for heart failure, non fatal myocardial infarction, and cardiac death.
Heart failure | 1 year.
  Heart failure (HF) is defined according to the diagnostic criteria for HF. Briefly, HF was defined as typical signs and symptoms of HF (NYHA class III or IV), as well as a history of myocardial infarct (MI) or with advanced coronary artery disease including severe 3-vessel disease and chronic total occlusion or other Organic heart disease.
Stroke | 1 year.
  Stroke was defined as a sudden onset of vertigo, numbness, aphasia, or dysarthria caused by cerebrovascular disease, including hemorrhage, embolism, thrombosis, or aneurysm rupture, and persisting for > 24 hours

SECONDARY OUTCOMES:
Main adverse cardiovascular and cerebrovascular events（MACCE） | 1 year.
  The composite endpoint for hospitalization for heart failure, non fatal myocardial infarction, cardiac death, and stroke.
Main adverse cardiovascular and cerebrovascular events（MACCE） | 3 years.
  The composite endpoint for hospitalization for heart failure, non fatal myocardial infarction, cardiac death, and stroke.
All cause death | 3 years.
  Death caused by various reasons.
Cardiac death | 3 years.
  Death caused by cardiac reasons.
Main adverse cardiovascular events（MACE） | 3 years.
  The composite endpoint for hospitalization for heart failure, non fatal myocardial infarction, and cardiac death.
Heart failure | 3 years.
  Heart failure (HF) is defined according to the diagnostic criteria for HF. Briefly, HF was defined as typical signs and symptoms of HF (NYHA class III or IV), as well as a history of myocardial infarct (MI) or with advanced coronary artery disease including severe 3-vessel disease and chronic total occlusion or other Organic heart disease.
Stroke | 3 years.
  Stroke was defined as a sudden onset of vertigo, numbness, aphasia, or dysarthria caused by cerebrovascular disease, including hemorrhage, embolism, thrombosis, or aneurysm rupture, and persisting for > 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Xie, Prof, Principal Investigator — Xinjiang Medical University
Locations (1):
- The First Affiliated Hospital of Xinjiang Medicial University, Ürümqi, Xinjiang, China

IPD SHARING:
Plan to Share IPD: Yes
Share the study protocol 6 months after the completion of the study.
Supporting Information: Study Protocol
Time Frame: 6 months after study completion.
Access Criteria: Sharing with scientific researchers.